CLINICAL TRIAL: NCT06281717
Title: A Pilot Study on the Role of Fetal Endotracheal Occlusion (FETO) in Fetuses with Severe Congenital Diaphragmatic Hernia
Brief Title: Fetal Endotracheal Occlusion (FETO) in Fetuses with Severe Congenital Diaphragmatic Hernia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alireza Shamshirsaz (Other)
Responsible Party: Sponsor-Investigator, Alireza Shamshirsaz, Director, Maternal Fetal Care Center, Boston Children's Hospital
Organization: Boston Children's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-P00045047
Record Dates: First submitted 2023-10-26; First posted 2024-02-28 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Congenital Diaphragmatic Hernia
Keywords: Hernias, Diaphragmatic, Congenital; Fetoscopic Endoluminal Tracheal Occlusion; Fetal Endoscopic Tracheal Occlusion; Hernia
MeSH Terms: conditions — Hernias, Diaphragmatic, Congenital; Hernia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Fetal Endotracheal Occlusion (FETO) (Experimental): Participants with severe congenital diaphragmatic hernia will undergo the FETO therapy.
  Interventions: Device: Fetal Endotracheal Occlusion (FETO)

INTERVENTIONS:
Device: Fetal Endotracheal Occlusion (FETO) — The FETO insertion procedure will be performed between gestational age 27 weeks 0 days and 29 weeks and 6 days. The Goldballoon Detachable Balloon (GOLDBAL2) will be inserted in the airway of the fetus using the Delivery Microcatheter (BALTACCI-BDPE100). The fetal tracheal balloon will be removed between 34 weeks 0 days and 34 weeks 6 days gestation or earlier as indicated.
  Other Names: Fetoscopic Endoluminal Tracheal Occlusion; FETO; Fetal Tracheal Occlusion; BALT GOLDBALLOON: GoldBAL2

SUMMARY:
The goal of this pilot trial is to learn more about the role of Fetal Endotracheal Occlusion (FETO) as an intervention in fetuses with severe congenital diaphragmatic hernia (CDH). The research team will investigate the feasibility and safety of the FETO procedure, as well as determine whether FETO can improve lung growth before birth, and survival after birth.

This study will enroll 10 pregnant participants to undergo the FETO procedure at a gestational age of 27 weeks 0 days to 29 weeks 6 days. The participant will be monitored for a few weeks, and then the FETO removal procedure will be performed ideally at 34 weeks 0 days to 34 weeks 6 days, but may be indicated earlier as determined by the Maternal Fetal care team. The pregnant participant and their baby will continue to be monitored during delivery and up until the child reaches 2 years of age.

DETAILED DESCRIPTION:
The goal of this study is to learn more about the role of Fetal Endotracheal Occlusion (FETO) as an intervention in fetuses with isolated severe congenital diaphragmatic hernia (CDH). CDH is a condition in which the diaphragm fails to completely close, leaving a gap through which abdominal organs can herniate and slide into and out of the chest. In severe cases, abdominal organs move into the chest and stay there, putting pressure on the heart and lungs and potentially causing the disruption or deformation of these structures. Impaired development of the lungs can often lead to a condition known as pulmonary hypertension, a form of high blood pressure that damages the heart. Pulmonary hypoplasia and pulmonary hypertension can be lethal. Congenital diaphragmatic hernia (CDH) affects 1 in 2,200 to 5,000 live births per year.

FETO will be performed with the goal of promoting lung growth and improving neonatal outcomes. FETO is a minimally invasive procedure in which a balloon device is inserted into the trachea of the fetus. The devices involved are the Goldballoon Detachable Balloon (GOLDBAL2) along with the Delivery Microcatheter (BALTACCI-BDPE100). The balloon would be left in place for several weeks and allow the lungs to grow, after which it would be removed, enabling the lungs to mature before birth. Participants will continue to be monitored up until the child reaches 2 years of age in order to assess mental and physical development after FETO.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patient 18 and older who is able to consent
* Singleton pregnancy
* Ability to reside within 30 minutes of Boston Children's Hospital for the duration of the FETO intervention, from the time of balloon placement until balloon removal
* Patient has a support person who is able to stay with them for the duration of the pregnancy

Fetal:

* Reassuring genetic analysis demonstrated by either normal Karyotype, normal fluorescence in situ hybridization (FISH) for chromosomes 13, 18, 21, X and Y, or chromosomal microarray (CMA) with non-pathologic variants
* Diagnosis of isolated left CDH with liver up
* Gestation at enrollment prior to 29 weeks 5 days
* SEVERE pulmonary hypoplasia with ultrasound Observed/Expected Lung-to-Head Ratio (O/E LHR) < 25%

Exclusion Criteria:

* Maternal contraindication to fetoscopic surgery or severe maternal medical condition in pregnancy
* Technical limitations precluding fetoscopic surgery, including uterine anomaly such as large or multiple fibroids, or Mullerian duct anomaly
* Latex allergy
* Preterm labor, shortened cervix (<20mm at enrollment or within 24 hours of FETO balloon insertion procedure) or uterine anomaly strongly predisposing to preterm labor, placenta previa
* Severe maternal obesity pre-pregnancy (BMI > 40)
* Psychosocial ineligibility, precluding consent, as determined by clinic social worker during review
* Inability to remain at FETO site during time period of tracheal occlusion, delivery, and postnatal care
* Right-sided or bilateral, left-sided CDH observed-to-expected lung to head ratio > 25% on ultrasound
* Additional fetal anomaly and chromosomal abnormalities by ultrasound, MRI, or echocardiogram that will significantly worsen prognosis
* History of incompetent cervix with or without cerclage
* Placental abnormalities (previa, abruption, accreta) known at time of enrollment
* Maternal-fetal RH (rhesus) isoimmunization, Kell sensitization, or neonatal alloimmune thrombocytopenia affecting the current pregnancy
* Maternal HIV, Hepatitis B, Hepatitis C status positive

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2031-02-28 (Estimated)

PRIMARY OUTCOMES:
Successful Ballon Placement | Gestational age of 27 weeks 0 days to 29 weeks 6 days
  Defined as direct visualization of balloon deployment above the carina at the time of FETO procedure
Successful Balloon Removal | Prior to delivery, ideally at 34 weeks
  Removal of the balloon prior to delivery, ideally during 34 weeks gestation
Balloon placement operative time | Gestational age of 27 weeks 0 days to 29 weeks 6 days
  Length of FETO procedure for successful balloon placement
Balloon removal operative time | Prior to delivery, ideally at 34 weeks
  Length of FETO procedure for successful balloon removal
Type of FETO release | Prior to delivery, ideally at 34 weeks
  Emergent or non-emergent FETO release
Maternal Complications | From balloon placement to delivery
  Maternal complications include: preterm labor, premature rupture of membranes, oligohydramnios, polyhydramnios, chorioamnionitis
Gestational age at delivery | At delivery
  Gestational age at delivery will be recorded

SECONDARY OUTCOMES:
Fetal lung volume | Once per week from balloon placement to removal. This measure will be recorded at earliest gestational age of 27 weeks 0 days, and latest at 34+6/7 weeks' gestation.
  Fetal lung volume will be monitored on ultrasound
Observed-to-Expected Lung to Head Ratio | Calculated at balloon removal, ideally at 34 weeks gestation
  Prenatal ultrasound will measure the observed-to-expected lung to head ratio (o/e LHR) at weekly visits while the balloon is in place and after balloon removal. Fetal lung growth will be calculated as the difference between the o/e LHR pre-balloon placement and the o/e LHR after balloon removal.
Infant survival | At hospital discharge or 6 months of age, whichever comes first. Hospital discharge typically occurs at 2-3 months of age
  Survival at discharge from the hospital, or at 6 months of age if still hospitalized
Oxygen dependency | At time of discharge, on average at 2-3 months of age
  Infant dependency on oxygen as defined by Bancalari 2001
Number of infants requiring ECMO (extracorporeal membrane oxygenation) | Birth to 6 months
  Use of ECMO support will be documented
NICU (neonatal intensive care unit) stay | From birth until discharge, at an average of 2-3 months of age
  Number of days spent in the neonatal intensive care unit
Ventilator support | Up to 2 years of age
  Number of days on ventilator support
Presence of periventricular leukomalacia | From birth until 2 months of age
  Incidence of periventricular leukomalacia at <2 months postnatally
Presence of neonatal sepsis | From birth until 1 month of age
  Incidence of neonatal sepsis
Presence of intraventricular hemorrhage | Up to 2 years of age
  Incidence of intraventricular hemorrhage (grade 0-III)
Retinopathy of prematurity | From birth to 1 month of age
  Incidence of retinopathy of prematurity (grade III or higher)
Presence of gastro-esophageal reflux | From birth until 2 years of age
  Incidence of gastro-esophageal reflux
CDH repair type | Postnatal, at time of CDH repair, typically within 2 weeks of birth
  CDH repair type will be documented as patch or muscle flap
Pulmonary function | At discharge around 2-3 months and at one year of age
  Pulmonary function by spirometry
Infant Neurodevelopment | At 6 months, 12 months, and 24 months of age
  Neurodevelopmental testing of the infant using the Bayley-4
Route of delivery | At delivery
  Delivery route will be recorded
Maternal hospitalization | From delivery until discharge, around 2-3 months of age
  Total days of maternal hospital stay after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Alireza Shamshirsaz, MD, Principal Investigator — Director, Maternal Fetal Care Center
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Done E, Gucciardo L, Van Mieghem T, Jani J, Cannie M, Van Schoubroeck D, Devlieger R, Catte LD, Klaritsch P, Mayer S, Beck V, Debeer A, Gratacos E, Nicolaides K, Deprest J. Prenatal diagnosis, prediction of outcome and in utero therapy of isolated congenital diaphragmatic hernia. Prenat Diagn. 2008 Jul;28(7):581-91. doi: 10.1002/pd.2033. PMID 18634116
- [Background] Deprest J, Jani J, Gratacos E, Vandecruys H, Naulaers G, Delgado J, Greenough A, Nicolaides K; FETO Task Group. Fetal intervention for congenital diaphragmatic hernia: the European experience. Semin Perinatol. 2005 Apr;29(2):94-103. doi: 10.1053/j.semperi.2005.04.006. PMID 16050527
- [Background] Saura L, Castanon M, Prat J, Albert A, Caceres F, Moreno J, Gratacos E. Impact of fetal intervention on postnatal management of congenital diaphragmatic hernia. Eur J Pediatr Surg. 2007 Dec;17(6):404-7. doi: 10.1055/s-2007-989275. PMID 18072025
- [Background] Deprest JA, Hyett JA, Flake AW, Nicolaides K, Gratacos E. Current controversies in prenatal diagnosis 4: Should fetal surgery be done in all cases of severe diaphragmatic hernia? Prenat Diagn. 2009 Jan;29(1):15-9. doi: 10.1002/pd.2108. No abstract available. PMID 19125386
- [Background] Harrison MR, Adzick NS, Estes JM, Howell LJ. A prospective study of the outcome for fetuses with diaphragmatic hernia. JAMA. 1994 Feb 2;271(5):382-4. PMID 8054005
- [Background] Metkus AP, Filly RA, Stringer MD, Harrison MR, Adzick NS. Sonographic predictors of survival in fetal diaphragmatic hernia. J Pediatr Surg. 1996 Jan;31(1):148-51; discussion 151-2. doi: 10.1016/s0022-3468(96)90338-3. PMID 8632269
- [Background] Keller RL, Glidden DV, Paek BW, Goldstein RB, Feldstein VA, Callen PW, Filly RA, Albanese CT. The lung-to-head ratio and fetoscopic temporary tracheal occlusion: prediction of survival in severe left congenital diaphragmatic hernia. Ultrasound Obstet Gynecol. 2003 Mar;21(3):244-9. doi: 10.1002/uog.44. PMID 12666218
- [Background] Albanese CT, Lopoo J, Goldstein RB, Filly RA, Feldstein VA, Calen PW, Jennings RW, Farrell JA, Harrison MR. Fetal liver position and perinatal outcome for congenital diaphragmatic hernia. Prenat Diagn. 1998 Nov;18(11):1138-42. doi: 10.1002/(sici)1097-0223(199811)18:113.0.co;2-a. PMID 9854721
- [Background] Stege G, Fenton A, Jaffray B. Nihilism in the 1990s: the true mortality of congenital diaphragmatic hernia. Pediatrics. 2003 Sep;112(3 Pt 1):532-5. doi: 10.1542/peds.112.3.532. PMID 12949279
- [Background] Does extracorporeal membrane oxygenation improve survival in neonates with congenital diaphragmatic hernia? The Congenital Diaphragmatic Hernia Study Group. J Pediatr Surg. 1999 May;34(5):720-4; discussion 724-5. doi: 10.1016/s0022-3468(99)90363-9. PMID 10359171
- [Background] Cacciari A, Ruggeri G, Mordenti M, Ceccarelli PL, Baccarini E, Pigna A, Gentili A. High-frequency oscillatory ventilation versus conventional mechanical ventilation in congenital diaphragmatic hernia. Eur J Pediatr Surg. 2001 Feb;11(1):3-7. doi: 10.1055/s-2001-12204. PMID 11370980
- [Background] Desfrere L, Jarreau PH, Dommergues M, Brunhes A, Hubert P, Nihoul-Fekete C, Mussat P, Moriette G. Impact of delayed repair and elective high-frequency oscillatory ventilation on survival of antenatally diagnosed congenital diaphragmatic hernia: first application of these strategies in the more "severe" subgroup of antenatally diagnosed newborns. Intensive Care Med. 2000 Jul;26(7):934-41. doi: 10.1007/s001340051284. PMID 10990109
- [Background] Muratore CS, Kharasch V, Lund DP, Sheils C, Friedman S, Brown C, Utter S, Jaksic T, Wilson JM. Pulmonary morbidity in 100 survivors of congenital diaphragmatic hernia monitored in a multidisciplinary clinic. J Pediatr Surg. 2001 Jan;36(1):133-40. doi: 10.1053/jpsu.2001.20031. PMID 11150452
- [Background] Muratore CS, Utter S, Jaksic T, Lund DP, Wilson JM. Nutritional morbidity in survivors of congenital diaphragmatic hernia. J Pediatr Surg. 2001 Aug;36(8):1171-6. doi: 10.1053/jpsu.2001.25746. PMID 11479850
- [Background] Boloker J, Bateman DA, Wung JT, Stolar CJ. Congenital diaphragmatic hernia in 120 infants treated consecutively with permissive hypercapnea/spontaneous respiration/elective repair. J Pediatr Surg. 2002 Mar;37(3):357-66. doi: 10.1053/jpsu.2002.30834. PMID 11877648
- [Background] Harrison MR, Jester JA, Ross NA. Correction of congenital diaphragmatic hernia in utero. I. The model: intrathoracic balloon produces fatal pulmonary hypoplasia. Surgery. 1980 Jul;88(1):174-82. PMID 7385020
- [Background] Harrison MR, Bressack MA, Churg AM, de Lorimier AA. Correction of congenital diaphragmatic hernia in utero. II. Simulated correction permits fetal lung growth with survival at birth. Surgery. 1980 Aug;88(2):260-8. PMID 6893089
- [Background] Harrison MR, Ross NA, de Lorimier AA. Correction of congenital diaphragmatic hernia in utero. III. Development of a successful surgical technique using abdominoplasty to avoid compromise of umbilical blood flow. J Pediatr Surg. 1981 Dec;16(6):934-42. doi: 10.1016/s0022-3468(81)80849-4. PMID 7200135
- [Background] Adzick NS, Outwater KM, Harrison MR, Davies P, Glick PL, deLorimier AA, Reid LM. Correction of congenital diaphragmatic hernia in utero. IV. An early gestational fetal lamb model for pulmonary vascular morphometric analysis. J Pediatr Surg. 1985 Dec;20(6):673-80. doi: 10.1016/s0022-3468(85)80022-1. PMID 4087097
- [Background] Harrison MR, Adzick NS, Longaker MT, Goldberg JD, Rosen MA, Filly RA, Evans MI, Golbus MS. Successful repair in utero of a fetal diaphragmatic hernia after removal of herniated viscera from the left thorax. N Engl J Med. 1990 May 31;322(22):1582-4. doi: 10.1056/NEJM199005313222207. No abstract available. PMID 2336088
- [Background] Harrison MR, Langer JC, Adzick NS, Golbus MS, Filly RA, Anderson RL, Rosen MA, Callen PW, Goldstein RB, deLorimier AA. Correction of congenital diaphragmatic hernia in utero, V. Initial clinical experience. J Pediatr Surg. 1990 Jan;25(1):47-55; discussion 56-7. doi: 10.1016/s0022-3468(05)80163-0. PMID 2405147
- [Background] Harrison MR, Adzick NS, Flake AW, Jennings RW, Estes JM, MacGillivray TE, Chueh JT, Goldberg JD, Filly RA, Goldstein RB, et al. Correction of congenital diaphragmatic hernia in utero: VI. Hard-earned lessons. J Pediatr Surg. 1993 Oct;28(10):1411-7; discussion 1417-8. doi: 10.1016/s0022-3468(05)80338-0. PMID 8263712
- [Background] Harrison MR, Adzick NS, Bullard KM, Farrell JA, Howell LJ, Rosen MA, Sola A, Goldberg JD, Filly RA. Correction of congenital diaphragmatic hernia in utero VII: a prospective trial. J Pediatr Surg. 1997 Nov;32(11):1637-42. doi: 10.1016/s0022-3468(97)90472-3. PMID 9396545
- [Background] Alcorn D, Adamson TM, Lambert TF, Maloney JE, Ritchie BC, Robinson PM. Morphological effects of chronic tracheal ligation and drainage in the fetal lamb lung. J Anat. 1977 Jul;123(Pt 3):649-60. PMID 885780
- [Background] Nardo L, Hooper SB, Harding R. Lung hypoplasia can be reversed by short-term obstruction of the trachea in fetal sheep. Pediatr Res. 1995 Nov;38(5):690-6. doi: 10.1203/00006450-199511000-00010. PMID 8552435
- [Background] Wilson JM, DiFiore JW, Peters CA. Experimental fetal tracheal ligation prevents the pulmonary hypoplasia associated with fetal nephrectomy: possible application for congenital diaphragmatic hernia. J Pediatr Surg. 1993 Nov;28(11):1433-9; discussion 1439-40. doi: 10.1016/0022-3468(93)90426-l. PMID 8301455
- [Background] DiFiore JW, Fauza DO, Slavin R, Peters CA, Fackler JC, Wilson JM. Experimental fetal tracheal ligation reverses the structural and physiological effects of pulmonary hypoplasia in congenital diaphragmatic hernia. J Pediatr Surg. 1994 Feb;29(2):248-56; discussion 256-7. doi: 10.1016/0022-3468(94)90328-x. PMID 8176601
- [Background] Hedrick MH, Estes JM, Sullivan KM, Bealer JF, Kitterman JA, Flake AW, Adzick NS, Harrison MR. Plug the lung until it grows (PLUG): a new method to treat congenital diaphragmatic hernia in utero. J Pediatr Surg. 1994 May;29(5):612-7. doi: 10.1016/0022-3468(94)90724-2. PMID 8035268
- [Background] Wild YK, Piasecki GJ, De Paepe ME, Luks FI. Short-term tracheal occlusion in fetal lambs with diaphragmatic hernia improves lung function, even in the absence of lung growth. J Pediatr Surg. 2000 May;35(5):775-9. doi: 10.1053/jpsu.2000.6067. PMID 10813348
- [Background] Luks FI, Wild YK, Piasecki GJ, De Paepe ME. Short-term tracheal occlusion corrects pulmonary vascular anomalies in the fetal lamb with diaphragmatic hernia. Surgery. 2000 Aug;128(2):266-72. doi: 10.1067/msy.2000.107373. PMID 10923003
- [Background] Flageole H, Evrard VA, Piedboeuf B, Laberge JM, Lerut TE, Deprest JA. The plug-unplug sequence: an important step to achieve type II pneumocyte maturation in the fetal lamb model. J Pediatr Surg. 1998 Feb;33(2):299-303. doi: 10.1016/s0022-3468(98)90451-1. PMID 9498406
- [Background] VanderWall KJ, Bruch SW, Meuli M, Kohl T, Szabo Z, Adzick NS, Harrison MR. Fetal endoscopic ('Fetendo') tracheal clip. J Pediatr Surg. 1996 Aug;31(8):1101-3; discussion 1103-4. doi: 10.1016/s0022-3468(96)90096-2. PMID 8863243
- [Background] VanderWall KJ, Skarsgard ED, Filly RA, Eckert J, Harrison MR. Fetendo-clip: a fetal endoscopic tracheal clip procedure in a human fetus. J Pediatr Surg. 1997 Jul;32(7):970-2. doi: 10.1016/s0022-3468(97)90379-1. PMID 9247214
- [Background] Harrison MR, Mychaliska GB, Albanese CT, Jennings RW, Farrell JA, Hawgood S, Sandberg P, Levine AH, Lobo E, Filly RA. Correction of congenital diaphragmatic hernia in utero IX: fetuses with poor prognosis (liver herniation and low lung-to-head ratio) can be saved by fetoscopic temporary tracheal occlusion. J Pediatr Surg. 1998 Jul;33(7):1017-22; discussion 1022-3. doi: 10.1016/s0022-3468(98)90524-3. PMID 9694087
- [Background] Flake AW, Crombleholme TM, Johnson MP, Howell LJ, Adzick NS. Treatment of severe congenital diaphragmatic hernia by fetal tracheal occlusion: clinical experience with fifteen cases. Am J Obstet Gynecol. 2000 Nov;183(5):1059-66. doi: 10.1067/mob.2000.108871. PMID 11084541
- [Background] Harrison MR, Sydorak RM, Farrell JA, Kitterman JA, Filly RA, Albanese CT. Fetoscopic temporary tracheal occlusion for congenital diaphragmatic hernia: prelude to a randomized, controlled trial. J Pediatr Surg. 2003 Jul;38(7):1012-20. doi: 10.1016/s0022-3468(03)00182-9. PMID 12861529
- [Background] Harrison MR, Albanese CT, Hawgood SB, Farmer DL, Farrell JA, Sandberg PL, Filly RA. Fetoscopic temporary tracheal occlusion by means of detachable balloon for congenital diaphragmatic hernia. Am J Obstet Gynecol. 2001 Sep;185(3):730-3. doi: 10.1067/mob.2001.117344. PMID 11568805
- [Background] Boland RE, Nardo L, Hooper SB. Cortisol pretreatment enhances the lung growth response to tracheal obstruction in fetal sheep. Am J Physiol. 1997 Dec;273(6):L1126-31. doi: 10.1152/ajplung.1997.273.6.L1126. PMID 9435566
- [Background] Ruano R, Peiro JL, da Silva MM, Campos JA, Carreras E, Tannuri U, Zugaib M. Early fetoscopic tracheal occlusion for extremely severe pulmonary hypoplasia in isolated congenital diaphragmatic hernia: preliminary results. Ultrasound Obstet Gynecol. 2013 Jul;42(1):70-6. doi: 10.1002/uog.12414. PMID 23349059
- [Background] Deprest JA, Benachi A, Gratacos E, Nicolaides KH, Berg C, Persico N, Belfort M, Gardener GJ, Ville Y, Johnson A, Morini F, Wielgos M, Van Calster B, DeKoninck PLJ; TOTAL Trial for Moderate Hypoplasia Investigators. Randomized Trial of Fetal Surgery for Moderate Left Diaphragmatic Hernia. N Engl J Med. 2021 Jul 8;385(2):119-129. doi: 10.1056/NEJMoa2026983. Epub 2021 Jun 8. PMID 34106555
- [Background] Deprest JA, Nicolaides KH, Benachi A, Gratacos E, Ryan G, Persico N, Sago H, Johnson A, Wielgos M, Berg C, Van Calster B, Russo FM; TOTAL Trial for Severe Hypoplasia Investigators. Randomized Trial of Fetal Surgery for Severe Left Diaphragmatic Hernia. N Engl J Med. 2021 Jul 8;385(2):107-118. doi: 10.1056/NEJMoa2027030. Epub 2021 Jun 8. PMID 34106556
- [Background] Van Calster B, Benachi A, Nicolaides KH, Gratacos E, Berg C, Persico N, Gardener GJ, Belfort M, Ville Y, Ryan G, Johnson A, Sago H, Kosinski P, Bagolan P, Van Mieghem T, DeKoninck PLJ, Russo FM, Hooper SB, Deprest JA. The randomized Tracheal Occlusion To Accelerate Lung growth (TOTAL)-trials on fetal surgery for congenital diaphragmatic hernia: reanalysis using pooled data. Am J Obstet Gynecol. 2022 Apr;226(4):560.e1-560.e24. doi: 10.1016/j.ajog.2021.11.1351. Epub 2021 Nov 19. PMID 34808130
- [Background] Jani JC, Nicolaides KH, Gratacos E, Valencia CM, Done E, Martinez JM, Gucciardo L, Cruz R, Deprest JA. Severe diaphragmatic hernia treated by fetal endoscopic tracheal occlusion. Ultrasound Obstet Gynecol. 2009 Sep;34(3):304-10. doi: 10.1002/uog.6450. PMID 19658113
- [Background] Jani JC, Nicolaides KH, Gratacos E, Vandecruys H, Deprest JA; FETO Task Group. Fetal lung-to-head ratio in the prediction of survival in severe left-sided diaphragmatic hernia treated by fetal endoscopic tracheal occlusion (FETO). Am J Obstet Gynecol. 2006 Dec;195(6):1646-50. doi: 10.1016/j.ajog.2006.04.004. Epub 2006 Jun 12. PMID 16769018
- [Background] Al-Maary J, Eastwood MP, Russo FM, Deprest JA, Keijzer R. Fetal Tracheal Occlusion for Severe Pulmonary Hypoplasia in Isolated Congenital Diaphragmatic Hernia: A Systematic Review and Meta-analysis of Survival. Ann Surg. 2016 Dec;264(6):929-933. doi: 10.1097/SLA.0000000000001675. PMID 26910202
- [Background] Ruano R, Lazar DA, Cass DL, Zamora IJ, Lee TC, Cassady CI, Mehollin-Ray A, Welty S, Fernandes CJ, Haeri S, Belfort MA, Olutoye OO. Fetal lung volume and quantification of liver herniation by magnetic resonance imaging in isolated congenital diaphragmatic hernia. Ultrasound Obstet Gynecol. 2014 Jun;43(6):662-9. doi: 10.1002/uog.13223. PMID 24127326
- [Background] Bebbington M, Victoria T, Danzer E, Moldenhauer J, Khalek N, Johnson M, Hedrick H, Adzick NS. Comparison of ultrasound and magnetic resonance imaging parameters in predicting survival in isolated left-sided congenital diaphragmatic hernia. Ultrasound Obstet Gynecol. 2014 Jun;43(6):670-4. doi: 10.1002/uog.13271. Epub 2014 May 5. PMID 24307080
- [Background] Perrone EE, Abbasi N, Cortes MS, Umar U, Ryan G, Johnson A, Ladino-Torres M, Ruano R; North American Fetal Therapy Network (NAFTNet). Prenatal assessment of congenital diaphragmatic hernia at north american fetal therapy network centers: A continued plea for standardization. Prenat Diagn. 2021 Jan;41(2):200-206. doi: 10.1002/pd.5859. Epub 2020 Nov 12. PMID 33125174
- [Background] Belfort MA, Olutoye OO, Cass DL, Olutoye OA, Cassady CI, Mehollin-Ray AR, Shamshirsaz AA, Cruz SM, Lee TC, Mann DG, Espinoza J, Welty SE, Fernandes CJ, Ruano R. Feasibility and Outcomes of Fetoscopic Tracheal Occlusion for Severe Left Diaphragmatic Hernia. Obstet Gynecol. 2017 Jan;129(1):20-29. doi: 10.1097/AOG.0000000000001749. PMID 27926636
- [Background] Baschat AA, Rosner M, Millard SE, Murphy JD, Blakemore KJ, Keiser AM, Kearney J, Bullard J, Nogee LM, Bembea M, Jelin EB, Miller JL. Single-Center Outcome of Fetoscopic Tracheal Balloon Occlusion for Severe Congenital Diaphragmatic Hernia. Obstet Gynecol. 2020 Mar;135(3):511-521. doi: 10.1097/AOG.0000000000003692. PMID 32028493
- [Background] Style CC, Olutoye OO, Belfort MA, Ayres NA, Cruz SM, Lau PE, Shamshirsaz AA, Lee TC, Olutoye OA, Fernandes CJ, Cortes MS, Keswani SG, Espinoza J. Fetal endoscopic tracheal occlusion reduces pulmonary hypertension in severe congenital diaphragmatic hernia. Ultrasound Obstet Gynecol. 2019 Dec;54(6):752-758. doi: 10.1002/uog.20216. Epub 2019 Nov 4. PMID 30640410
- [Background] Donepudi R, Belfort MA, Shamshirsaz AA, Lee TC, Keswani SG, King A, Ayres NA, Fernandes CJ, Sanz-Cortes M, Nassr AA, Espinoza AF, Style CC, Espinoza J. Fetal endoscopic tracheal occlusion and pulmonary hypertension in moderate congenital diaphragmatic hernia. J Matern Fetal Neonatal Med. 2022 Dec;35(25):6967-6972. doi: 10.1080/14767058.2021.1932806. Epub 2021 Jun 6. PMID 34096456
- [Background] Russo FM, Cordier AG, Basurto D, Salazar L, Litwinska E, Gomez O, Debeer A, Nevoux J, Patel S, Lewi L, Pertierra A, Aertsen M, Gratacos E, Nicolaides KH, Benachi A, Deprest J. Fetal endoscopic tracheal occlusion reverses the natural history of right-sided congenital diaphragmatic hernia: European multicenter experience. Ultrasound Obstet Gynecol. 2021 Mar;57(3):378-385. doi: 10.1002/uog.23115. PMID 32924187
- [Background] Espinoza J, King A, Shamshirsaz AA, Nassr AA, Donepudi R, Sanz Cortes M, Meholin-Ray AR, Krispin E, Johnson R, Mendez Martinez Y, Keswani SG, Lee TC, Joyeux L, Espinoza AF, Olutoye Ii O, Garcia-Prats JA, Fernandes CJ, Coleman RD, Lohmann P, Rhee CJ, Davies J, Belfort MA. Characterization of Suboptimal Responses to Fetoscopic Endoluminal Tracheal Occlusion in Congenital Diaphragmatic Hernia. Fetal Diagn Ther. 2023;50(2):128-135. doi: 10.1159/000530549. Epub 2023 Apr 11. PMID 37040717
- [Background] Fallon SC, Cass DL, Olutoye OO, Zamora IJ, Lazar DA, Larimer EL, Welty SE, Moise AA, Demny AB, Lee TC. Repair of congenital diaphragmatic hernias on Extracorporeal Membrane Oxygenation (ECMO): does early repair improve patient survival? J Pediatr Surg. 2013 Jun;48(6):1172-6. doi: 10.1016/j.jpedsurg.2013.03.008. PMID 23845603
- [Background] Vergote S, De Bie FR, Duffy JMN, Bosteels J, Benachi A, Power B, Meijer F, Hedrick HL, Fernandes CJ, Reiss IKM, De Coppi P, Lally KP, Deprest JA. Core outcome set for perinatal interventions for congenital diaphragmatic hernia. Ultrasound Obstet Gynecol. 2023 Sep;62(3):374-382. doi: 10.1002/uog.26235. Epub 2023 Aug 7. PMID 37099763